CLINICAL TRIAL: NCT07109050
Title: The Effectiveness of Virtual Reality Interventions Within Specialist Palliative Care (VR-SPC): A Hermeneutic Single Case Efficacy Design (HSCED) Series
Brief Title: Virtual Reality Within Palliative Care (VR-SPC)
Acronym: VR-SPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lincoln (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 349429
Record Dates: First submitted 2025-07-21; First posted 2025-08-07 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Palliative Care; Virtual Reality; Wellbeing
Keywords: virtual reality; palliative care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention - VR (Other): Participants will be offered a VR intervention, whereby they will decide what VR experience they would like to use, picked from a pre-set list. VR experiences will be picked inline with pre-determined goals set by participants in the initial session of the study. VR expereinces range from ocean views, city experiences, to animals.
  Interventions: Device: VR Headset

INTERVENTIONS:
Device: VR Headset — VR will be offered on either an individual or joint-experience basis, whereby the participant(s) wear a VR headset with 360 degree views, to explore various VR experiences of their choice for up to 3 sessions on a weekly basis. Goals for using VR will be ascertained by completing the goal based measure with the patient who is accessing specialist palliative care. This will define the purpose of the VR intervention in future sessions. The participant will be shown a list of VR experience options so they are aware of these prior to the next session. Pre-VR and post-VR questionnaires will be completed.
  Other Names: VR

SUMMARY:
Literature so far shows VR is largely acceptable and feasible to use in palliative care settings, especially for improving patient wellbeing and mental health. However, limited research exists for understanding the effectiveness of VR, especially if sessions are repeated or offered jointly with patient carers or companions. We aim to investigate the effectiveness of VR for achieving personally meaningful goals (including but not limited to relaxation, bucket-list activities, and improving wellbeing). This study will be offered to patients and their companions receiving palliative care at a hospice in England. Informed consent will be acquired after a participant information sheet has been shared with interested participants. Personal goals of VR use will be established at the start of the study with baseline mental health and wellbeing data collection. Up to 3 VR sessions will be offered.

Before and after each session patients will be asked to complete questionnaires to track wellbeing and progression towards intended goals for utilising VR. A change interview will occur between 1 to 4 weeks after the final VR session to discuss their overall experiences of VR and will include repeated follow up questionnaires. Participants that which to engage with a joint-VR intervention with their companion (referred to as participant companions for the purposes of this study), will also require informed consent and completion of questionnaires and interview attendance to be involved with this study.

Results will be gathered and analysed by creating anonymous individual rich case records and shared with a panel of independent psychologists to conclude whether or not, from our findings, virtual reality is effective for achieving personally important goals. Findings will be shared with the hospice involved and form a Doctoral Thesis based at the University of Lincoln.

DETAILED DESCRIPTION:
Patients who are accessing palliative care have progressive or terminal illness. Patients may also have co-occurring mental health difficulties or reduced wellbeing. There is emerging evidence for psychological wellbeing benefits of non-pharmacological interventions in palliative care. Also it is important for patient's receiving palliative care to have autonomy, dignity and respect in the care they receive (see Ambitions for Palliative and End of Life Care: A national framework for local action 2021-2026). One way to achieve such ambitions and offer an intervention for wellbeing is that of Virtual Reality (VR), whereby an individual is immersed in a digital world by wearing a headset. Immersive experiences can provide patients with a sense of being somewhere new which they may not be able to physically reach due to a decline in health or mobility inline with their palliative needs (Altman et al., 2024).

This study adopts a hermeneutic single case efficacy design (HSCED)series, which involves creating case studies that track up to 6 participants taking part in a 4-week VR intervention. The intervention offered for the study will be psychologically informed in that VR experiences and purpose for the intervention use will be chosen by the patient inline with their own personally important and meaningful goals. By ensuring that choice of the VR intervention offered will promote self-determination in care (e.g. autonomy and relatedness). While also acknowledging patient companion's experiences if patients choose to use VR jointly with their family member or companion, patient companions would also be interviewed about their experience of using VR.

Mixed-methods data collection will occur including quantitative data (questionnaires, number of sessions, time spent wearing VR) and qualitative data (interviews will occur to understand participant experience of using VR). Overall, this study will add to current literature about the effectiveness of VR for patients in palliative care.

ELIGIBILITY:
Inclusion criteria:

Participants recieving palliative care must be:

* Aged 18 or over (no upper age limit due to the service being lifelong).
* Patients deemed to be palliative, receiving specialist care at the designated hospice as either an inpatient or outpatient.
* Willing and able to engage in VR interventions as determined by the patients' usual care team.
* Able to consent to the research, as assessed by the clinical psychologist supporting recruitment and the primary researcher delivering the VR intervention.

Participant companions (carers, relatives) must be:

* Aged 18 or over (no upper age limit).
* Willing and able to engage in VR interventions and travel to the designated hospice site.
* Able to consent to the research, as assessed by the clinical psychologist supporting recruitment and the primary researcher delivering the VR intervention.

Exclusion criteria:

* Lacking capacity to consent to take part in research as assessed by both the clinical psychologist supporting recruitment and the primary researcher delivering VR.
* Exhibiting contraindications as set out by care team including eyesight impairments or neurological conditions such as epilepsy or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-4; Kroeneke et al., 2009) | Baseline, week 1, week 2, week 3, and at week 8 (follow up interview).
  Depression and anxiety measure. 4 items. 4-point Likert Scale (0 = Not at all, 3 = Nearly every day). Wording of the question and options will be adapted for post-VR use to include 'how much are you feeling bothered by the following problems now?' along with options changed to 'not at all', 'a little bit', 'somewhat', 'a lot'. Higher scores indicate higher likelihood of depression and anxiety, whereby:
  * None = 0-2
  * Mild = 3-5
  * Moderate = 6-8
  * Severe = 9-12 On each subscale, a score of 3 or greater is considered positive for screening purposes.
The Functional Assessment of Chronic Illness Therapy-Palliative (FACIT-Pal) 14 (FACIT PAL-14; Zeng et al., 2013). | Baseline and week 8 (follow up interview).
  Quality of life measure for palliative care patients. 14 items. 5-point Likert Scale (0 = Not at all, 5 = Very much). Higher score indicates a better quality of life.
Edmonton Symptom Assessment Scale (ESAS; Bruera et al., 1991) | Baseline and week 8 (follow up interview).
  Assesses pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, and shortness of breath. 10 items. Each symptom is rated on a scale of 0 (no symptom) to 10 (worst possible symptom). Higher scores indicate higher incidents and severity of symptoms.
• Goal based outcome measures (GBO; Law & Jacob, 2015) | Baseline, week 1, week 2, and week 3.
  To set individual goals for interventions and track progress. Up to 3 goals set, and tracking on a scale from 0 to 10 how much an individual feels they are achieving their goal. Progress is monitored overtime.
Change interview procedure based on the 'Change interview' (Elliot et al., 1999) | Week 8 (follow up interview).
  Interview to understand individual changes since VR intervention, as well as helpful and unhelpful aspects of an intervention, what has brought change. To be used as a guide and to inspire interviewer prompts.

SECONDARY OUTCOMES:
Non validated - Rating scale to assess subjective ratings of VR experience | Week 1, week 2, and week 3.
  How immersed into the VR experience did you feel on a scale of 1 to 10 where 0 = not immersed at all, 10 = fully immersed? The wording of this question may differ depending on the VR experience selected, such as "how much did you feel like you were swimming with the dolphins, with 1 being not at all, and 10 being like you were right there with the dolphins?" to aid understanding of the question
Helpful Aspects of Therapy (HAT; Llewelyn, 1988) | Week 1, week 2, and week 3.
  To understand helpful and unhelpful aspects of an intervention. 7 items. Open-ended questions whereby participants describe in their own words the most helpful and unhelpful aspects of the session. Wording will be adapted for the purposes of this study to apply to VR sessions as opposed to 'therapy'.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lincoln, Lincoln, United Kingdom

IPD SHARING:
Plan to Share IPD: No
To protect participant confidentiality due to sensitive nature of the palliative care setting.